CLINICAL TRIAL: NCT05402462
Title: Esophageal Motility Disorders in Patients With Non-cardiac Chest Pain at Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa medhat Ahmed, principal Investigator, Assiut University
Other Study IDs: Esophageal motility disorders
Record Dates: First submitted 2022-02-18; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-02

CONDITIONS: Esophageal Motility Disorders
MeSH Terms: conditions — Esophageal Motility Disorders | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: upper endoscopy — detect esphageal motility disorder by upper endoscopy and esophageal manometry
  Other Names: esophageal manometry

SUMMARY:
to determine the prevalence and distribution of esophageal motility disorders in NCCP patients who presented after a negative cardiac evaluation and underwent esophageal manometry, esophageal pH monitoring

DETAILED DESCRIPTION:
Non-cardiac chest pain (NCCP) is defined as recurrent anginalike pain without evidence of cardiac disease [1]. NCCP is a common disorder and accounts for 14-33% of patient visits to gastroenterologists [2]. These patients frequently undergo testing for reflux and esophageal motility as gastroesophageal reflux disease (GERD) is seen in 50-60% and esophageal motility disorders in 15-18% of the patients [3,4]. Nutcracker esophagus was thought to be the classic manometric finding in NCCP [5] but other studies have reported ineffective esophageal motility (IEM) as the most common motility disorder in NCCP [6,7]. Furthermore, up to one-third of patients do not have any GERD or motility disorders and are labeled as functional chest pain [8]. Suggested causes in these patients include esophageal hypersensitivity [9], abnormal cerebral pain processing and psychological comorbidity [10]. The clinical predictors of abnormal esophageal function tests in NCCP have not been identified. Identifying these factors would lead to limited use of testing in those with risk factors and faster institution of pain modulator therapy in patients who are most likely to have functional chest pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Patients presented with non-cardiac chest pain

Exclusion Criteria:

* 1- age below 18. 2- cardiac chest pain patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: to determine the prevalence and distribution of esophageal motility disorders in NCCP patients who presented after a negative cardiac evaluation and underwent esophageal manometry, esophageal pH monitoring
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Esophageal motility disorders in patients with non-cardiac chest pain at Assiut University hospital | one year
  Determine esophageal motility disorder in patient with non cardiac chest pain using ECG ,cardiac enzymes and echocardiography , esophageal manometry and upper endoscopy

REFERENCES:
- [Result] Fass R, Achem SR. Noncardiac chest pain: epidemiology, natural course and pathogenesis. J Neurogastroenterol Motil. 2011 Apr;17(2):110-23. doi: 10.5056/jnm.2011.17.2.110. Epub 2011 Apr 27. PMID 21602987
- [Result] Yamasaki T, Fass R. Noncardiac chest pain: diagnosis and management. Curr Opin Gastroenterol. 2017 Jul;33(4):293-300. doi: 10.1097/MOG.0000000000000374. PMID 28463855
- [Result] Coss-Adame E, Rao SS. A Review of Esophageal Chest Pain. Gastroenterol Hepatol (N Y). 2015 Nov;11(11):759-66. PMID 27134590
- [Result] Fass R, Dickman R. Non-cardiac chest pain: an update. Neurogastroenterol Motil. 2006 Jun;18(6):408-17. doi: 10.1111/j.1365-2982.2006.00787.x. PMID 16700719
- [Result] Katz PO, Dalton CB, Richter JE, Wu WC, Castell DO. Esophageal testing of patients with noncardiac chest pain or dysphagia. Results of three years' experience with 1161 patients. Ann Intern Med. 1987 Apr;106(4):593-7. doi: 10.7326/0003-4819-106-4-593. PMID 3826958
- [Result] Ribolsi M, Balestrieri P, Biasutto D, Emerenziani S, Cicala M. Role of Mixed Reflux and Hypomotility with Delayed Reflux Clearance in Patients with Non-cardiac Chest Pain. J Neurogastroenterol Motil. 2016 Oct 30;22(4):606-612. doi: 10.5056/jnm15182. PMID 27095707
- [Result] Barret M, Herregods TV, Oors JM, Smout AJ, Bredenoord AJ. Diagnostic yield of 24-hour esophageal manometry in non-cardiac chest pain. Neurogastroenterol Motil. 2016 Aug;28(8):1186-93. doi: 10.1111/nmo.12818. Epub 2016 Mar 27. PMID 27018150
- [Result] Remes-Troche JM. How to Diagnose and Treat Functional Chest Pain. Curr Treat Options Gastroenterol. 2016 Dec;14(4):429-443. doi: 10.1007/s11938-016-0106-y. PMID 27709331
- [Result] Farmer AD, Ruffle JK, Aziz Q. The Role of Esophageal Hypersensitivity in Functional Esophageal Disorders. J Clin Gastroenterol. 2017 Feb;51(2):91-99. doi: 10.1097/MCG.0000000000000757. PMID 28005634
- [Result] Zhang L, Tu L, Chen J, Song J, Bai T, Xiang XL, Wang RY, Hou XH. Health-related quality of life in gastroesophageal reflux patients with noncardiac chest pain: Emphasis on the role of psychological distress. World J Gastroenterol. 2017 Jan 7;23(1):127-134. doi: 10.3748/wjg.v23.i1.127. PMID 28104988